CLINICAL TRIAL: NCT05220098
Title: A Phase 1/2, First-in-Human, Open-Label, Dose-Escalation Study of TAK-280 in Patients With Unresectable Locally Advanced or Metastatic Cancer
Brief Title: First-in-Human Study of TAK-280 in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to limited anti-cancer activity
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-280-1501; 2023-504012-16-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2022-01-07; First posted 2022-02-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Unresectable Locally Advanced or Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Dose-escalation Phase is non-randomized and Cohort-expansion Phase will include randomized and non-randomized cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose-escalation Phase: TAK-280 (Experimental): Participants will receive TAK-280 intravenous (IV) infusion on Days 1, 8, 15, and 22 of a 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal from study occurs.
  Interventions: Drug: TAK-280
- Cohort-expansion Phase: TAK-280 High or low Dose (Experimental): Participants will receive either TAK-280 high or low dose in one selected indication and only one dose level of TAK-280 in the remaining indications as determined from the dose-escalation phase of the study in 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal from study occurs.
  Interventions: Drug: TAK-280

INTERVENTIONS:
Drug: TAK-280 — Participants will receive TAK-280 as IV infusion.

SUMMARY:
The main aim of this study is to find out the safety, tolerability, and effect of TAK- 280 in participants with unresectable, locally advanced or metastatic cancer who have experienced treatment failure or are intolerant to standard therapies.

Participants will be treated with TAK-280 for up to 14 treatment cycles. Each treatment cycle will be 28 days.

After the last dose of study drug, participants will be followed up for survival every 12 weeks for a total of 48 weeks.

DETAILED DESCRIPTION:
This study consists of 2 phases: Dose-escalation and cohort-expansion phase.

Dose-escalation phase:

The purpose of the dose-escalation phase is to generate data to characterize the initial safety and tolerability profile of TAK-280 and determine the 2 recommended doses for expansion (RDEs) of TAK-280 to be administered during the cohort-expansion phase.

Cohort-Expansion Phase:

The cohort expansion phase will be conducted in 3 indications. Only in 1 selected indication participants will be randomized 1:1 to receive either TAK-280 high dose or low dose. In the remaining 2 indications to be studied in the cohort-expansion phase, participants will receive only one dose level of TAK-280.

ELIGIBILITY:
Inclusion Criteria

* Age greater than or equal to (>=)18 years or >= the local legal age of majority, as applicable.
* Criteria for disease state in dose escalation and cohort expansion.

  1. Tumor histologies during dose escalation: Dose escalation will begin by initially enrolling participants with histologically or pathologically confirmed, unresectable, locally advanced or metastatic cancers.
  2. Tumor histologies during cohort expansion: Participants will be eligible if they have histologically proven, unresectable, locally advanced or metastatic malignant neoplasms.
* Eastern Cooperative Oncology Group performance status (less than or equal to [<=]) 1.
* Measurable disease per RECIST V1.1 by investigator except for participants with mCRPC with bone metastases only (these participants are allowed in the study). Lesions in previously irradiated areas (or other local therapy) should not be selected as measurable/target lesions, unless treatment was >=6 months prior to start of treatment or there has been demonstrated progression with a clear margin to measure in that particular lesion.

Exclusion Criteria

* History of known autoimmune disease.
* Major surgery or traumatic injury within 8 weeks before the first dose of TAK-280.
* Unhealed wounds from surgery or injury.
* Ongoing or active infection of Grade >=2.
* Oxygen saturation less than (<) 92 percent (%) on room air at screening or during Cycle 1 Day 1 (C1D1) predose assessment.
* Inflammatory process that has not resolved for >= 4 weeks before the first dose of study drug. Participants with chronic low-grade inflammatory processes such as radiation-induced pneumonitis are excluded regardless of their duration.
* Vaccination with any live virus vaccine within 4 weeks or other vaccines within 2 weeks before the initiation of study drug administration. Inactivated annual influenza vaccination is allowed.
* Known hypersensitivity to TAK-280 or any excipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | From start of the initial dose up to Cycle 1 Day 28
  DLT evaluation period is defined as the time between the initial dose of TAK-280 and Cycle 1 Day 28.
Number of Participants With Treatment- emergent Adverse Events (TEAEs) | Up to approximately 37 months

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of TAK-280 | Pre-dose and at multiple time points post-dose on Days 1, 2, 3, 8, 15, 22 up to the end of treatment (Up to 14 months)
  Cmax of TAK-280 will be reported.
Area Under Plasma Concentration-Time Curve (AUC) of TAK- 280 | Pre-dose and at multiple time points post-dose on Days 1, 2, 3, 8, 15, 22 up to the end of treatment (Up to 14 months)
  AUC of TAK-280 will be reported.
Time to Reach Maximum Observed Plasma Concentration (tmax) of TAK-280 | Pre-dose and at multiple time points post-dose on Days 1, 2, 3, 8, 15, 22 up to the end of treatment (Up to 14 months)
  tmax of TAK-280 will be reported.
Terminal Disposition Phase Half-Life (t1/2) of TAK-280 | Pre-dose and at multiple time points post-dose on Days 1, 2, 3, 8, 15, 22 up to the end of treatment (Up to 14 months)
  t1/2 of TAK-280 will be reported.
Total Clearance (CL) of TAK-280 | Pre-dose and at multiple time points post-dose on Days 1, 2, 3, 8, 15, 22 up to the end of treatment (Up to 14 months)
  CL of TAK-280 will be reported.
Volume of Distribution at Steady State (Vss) After IV Administration of TAK-280 | Pre-dose and at multiple time points post-dose on Days 1, 2, 3, 8, 15, 22 up to the end of treatment (Up to 14 months)
  Vss of TAK-280 will be reported.
Confirmed Overall Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST V1.1) | Up to approximately 37 months
  ORR is defined as the percentage of participants who achieve confirmed complete response (CR) or partial response (PR) based on RECIST V1.1 as determined by the investigator during the study.
Duration of Response (DOR) Based on RECIST V1.1 | Up to approximately 37 months
  DOR is defined as the time from the date of first documentation of a PR or better to the date of first documentation of progressive disease (PD) or death due to any cause, whichever occurs first, for participants with a confirmed response (PR or better).
Progression Free Survival (PFS) | From start of first dose to disease progression or death, whichever occurred first (up to approximately 37 months)
  PFS is defined as the time from the date of the first dose of TAK-280 to the date of first documentation of PD or death due to any cause, whichever occurs first.
Overall Survival (OS) | From start of first dose of study drug up to death (up to approximately 37 months)
  OS is defined as the time from the date of the first dose of TAK-280 to the date of death due to any cause.
Disease Control Rate | Up to approximately 37 months
  Disease control rate is defined as the percentage of participants who achieve PR or CR or SD, with a duration of greater than or equal to (>=) 2 consecutive scans.
Percentage of Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) Having Prostate-Specific Antigen (PSA) Response | Up to approximately 37 months
  PSA response is defined as PSA reduction from baseline of >= 50 percent (%) and confirmed at least 3 weeks later.
Duration of PSA Response in Participants With mCRPC | Up to approximately 37 months
  Duration of PSA response is defined as the time from first PSA response to first documented PSA progression.
Time to PSA Progression in Participants With mCRPC | Up to approximately 37 months
  Time to PSA progression is defined as the time from the date of first dose of TAK-280 to the date that an increase of 25% or more and absolute increase of 2 nanograms/milliliter (ng/mL) or more from the nadir.
Percentage of Participants With mCRPC Having PSA Reductions of >= 50% up to 6 Months | Baseline up to 6 months
Percentage of Participants who Develop Positive Induced Antidrug Antibody (ADA) for TAK-280 | Cycle 1 to 5: pre-dose (Each cycle= 28 days)
Percentage of Participants who Developed Neutralizing Antibody (NAb) Titers for TAK-280 | Cycle 1 to 5: pre-dose (Each cycle= 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- United States (10):
  - University of Arkansas For Medical Sciences, Little Rock, Arkansas
  - University of California San Francisco, San Francisco, California
  - University of Minnesota - Masonic Cancer Center, Minneapolis, Minnesota
  - Duke Cancer Institute, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - SCRI Tennessee Oncology Nashville, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Chris O'Brien Lifehouse Hospital, Camperdown, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park
  - Monash Medical Centre, Clayton
  - Cabrini Health, Malvern
- Canada (2):
  - Centre Intégré de Cancérologie du CHU de Québec - Université Laval, Québec
  - Centre Hospitalier Universitaire de Sherbrooke CHUS, Sherbrooke
- Spain (7):
  - Hospital Quironsalud Barcelona, NEXT Oncology, Barcelona
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Instituto de Investigacion Oncologica Vall dHebron (VHIO) - EPON, Barcelona
  - START MADRID_Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/dbc0aa0e1b69463d?idFilter=%5B%22TAK-280-1501%22%5D